CLINICAL TRIAL: NCT05869682
Title: Phase 2 Study of Bright White Light During Treatment With ADT Combination Therapy in Men With Advanced Prostate Cancer to PreServe PHysIcal and MeNtal HEalth (SHINE)
Brief Title: Bright White Light Therapy in Reducing Cancer-Related Fatigue and Depression in Advanced Prostate Cancer Patients Undergoing Treatment With ADT Combination Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22628; NCI-2023-03486 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22628 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Advanced Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Carcinoma; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultraviolet Therapy; Drug Therapy, Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, only the designated study team member knows the participant's allocation. Oncologists or clinical research associates collecting data are not informed of patient allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group I (Immediate BWL therapy) (Experimental): Patients wear AYOpro BWL therapy glasses starting on day 1 of SOC ADT combination therapy for 12 months on trial.
  Interventions: Procedure: Bright White Light Therapy; Drug: Combination Drug Therapy; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Group II (Delayed BWL therapy) (Experimental): Patients wear AYOpro BWL therapy glasses starting 6 months after the start of SOC ADT combination therapy for 6 months on trial.
  Interventions: Procedure: Bright White Light Therapy; Drug: Combination Drug Therapy; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Bright White Light Therapy — Wear AYOpro BWL therapy
  Other Names: Bright Light Therapy; Bright White Light; BWL
Drug: Combination Drug Therapy — Receive SOC ADT combination therapy
  Other Names: Drug Therapy, Combination
Other: Electronic Health Record Review — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Group II (Delayed BWL therapy)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well bright white light (BWL) therapy works in reducing cancer-related fatigue and depression in patients with prostate cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and who are undergoing treatment with antiandrogen therapy (ADT) combination therapy. Combination treatment including ADT plus chemotherapy and androgen receptor (AR) targeted therapy or ADT plus AR targeted therapies work by reducing testosterone. Most prostate tumor cells rely on testosterone to help them grow; therefore, ADT combination therapy causes prostate tumor cells to die or to grow more slowly leading to improved overall survival in men with advanced prostate cancer when compared with ADT alone. However, lower levels of testosterone is also commonly associated with worsening fatigue and depression. If prolonged and severe, these complications can alter patient treatment plans, impacting not just quality of life, but leading to inadequate cancer control. BWL therapy is a type of phototherapy that utilizes bright white full-spectrum light, either through a light box or light therapy glasses to help regulate circadian rhythms. Circadian rhythms are physical, mental, and behavioral changes that follow a 24-hour cycle, including the sleep-wake cycle which can become disrupted in cancer patients undergoing treatment, leading to increased fatigue. Additionally, exposure to bright light may increase the production of serotonin, a neurotransmitter that is associated with mood regulation. BWL therapy with AYOpro light therapy glasses may serve as a supportive care measure for men with advanced prostate to help reduce fatigue, as well as improve mood and overall quality of life during ADT combination therapy to maintain cancer care without suffering complications of therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether patient-reported fatigue by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue instrument at 3 months is lower in men with prostate cancer receiving immediate bright white light therapy as compared with delayed bright white light (BWL) therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT+ hormonal intensification).

SECONDARY OBJECTIVES:

I. To evaluate the difference in the following outcomes between men with prostate cancer receiving immediate bright white light therapy as compared with delayed bright white light (BWL) therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT + hormonal intensification):

Ia. Mood by the Patient Health Questionnaire (PHQ)-9 instrument measuring depressive symptoms; Ib. Geriatric assessments by the Cancer and Aging Research Group- Geriatric Assessment (CARG-GA) and Geriatric 8 (G8) instruments; Ic. Overall quality of life by the Functional Assessment of Cancer Therapy (FACT)-Prostate (FACT-P) instrument.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (IMMEDIATE): Patients wear AYOpro BWL therapy glasses starting on day 1 of standard of care (SOC) ADT combination therapy for 12 months on trial.

GROUP II (DELAYED): Patients wear AYOpro BWL therapy glasses starting 6 months after the start of SOC ADT combination therapy for 6 months on trial.

Patients are followed for 52 weeks (total duration of the trial), or for 4 weeks including after removal from protocol therapy or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer
* Participants must have radiographic evidence of measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 10 mm ( >= 1 cm) with computed tomography (CT) scan or magnetic resonance imaging (MRI), or metastatic lesions as identified as related to prostate cancer on a standard technetium bone scan. Alternatively patients may have radiographic evidence of metastatic disease on an Axumin or prostate-specific membrane antigen (PSMA)-positron emission tomography (PET) scan
* Eligible for treatment with ADT plus docetaxel (planned for 6 cycles or fewer) plus abiraterone acetate and prednisone or darolutamide (triplet therapy), or ADT plus enzalutamide, apalutamide, or darolutamide (doublet therapy). Prior use of ADT with a gonadotropin hormone-releasing hormone (GnRH) agonist or antagonist, or prior orchiectomy is allowed
* Age >= 60 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Expected time to next treatment of >= 12 months and life expectancy of >= 18 months, as determined by a study Investigator
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< institutional ULN OR
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better
* Ability to understand and the willingness to sign a written informed consent document
* Participants are still eligible and may proceed with the protocol and bright white light therapy if they discontinue baseline hormonal treatment, but plan to continue with another of the eligible treatments. However, if they discontinue treatment due to cancer progression, they should not continue on the protocol

Exclusion Criteria:

* Participants receiving docetaxel cannot have metastatic castration-resistant prostate cancer as the expected median time to progression to next therapy is < 12 months
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Prior treatment with combination hormonal therapy with abiraterone acetate, enzalutamide, apalutamide, or darolutamide for participants planning to start treatment with abiraterone acetate, enzalutamide, apalutamide, or darolutamide
* Participants who are receiving any other investigational agents
* Participants with brain metastases are ineligible due to the limited life expectancy of men with prostate cancer metastases to brain
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study
* Histologic evidence of small cell prostate cancer
* Symptomatic skeletal event complication of prostate cancer such as cord compression, fracture, or need for radiation or surgery to a bone lesion within 6 months
* Uncontrolled pain related to prostate cancer or separate chronic condition
* Visceral crisis from prostate cancer suggesting rapidly progressive disease and life expectancy of < 18 months
* Participants with uncontrolled intercurrent illness
* Concurrent second active malignancy
* Severe sleep disorders (e.g. Narcolepsy)
* Eye Diseases which limit the ability of light to be processed (e.g. untreated cataracts, severe glaucoma, macular degeneration, blindness, pupil dilation problems or other retinal disorder)
* Severe psychological impairment (e.g., bipolar disorder or manic episodes)
* Current employment in night shift work
* Previous use of light therapy to alleviate fatigue or depressive symptoms
* Currently recovering from previous eye surgery within the past 6 months that causes eye irritation
* Sensitivity to light, epilepsy, or a history of seizures

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported fatigue | Baseline to 3 months post antiandrogen therapy (ADT) combination treatment initiation
  Will compare patient-reported fatigue between men treated with immediate versus delayed bright white light (BWL) therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT+ hormonal intensification). Measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue instrument. T test will be used to compare FACIT-Fatigue change score between two arms (T2 [3 month after treatment initiation] minus T1 [before or at treatment initiation]).

SECONDARY OUTCOMES:
Difference in mood outcomes | Baseline to 3 months post ADT combination treatment initiation
  Will compare the difference in mood between men with prostate cancer receiving immediate BWL therapy as compared with delayed BWL therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT + hormonal intensification). Measured by Patient Health Questionnaire (PHQ)-9 instrument measuring depressive symptoms. T test will be used to compare PHQ-9 change score between two arms (T2 [3 month after treatment initiation] minus T1 [before or at treatment initiation]).
Difference in geriatric assessments | Baseline to 3 months post ADT combination treatment initiation
  Will compare the difference in geriatric assessments between men with prostate cancer receiving immediate BWL therapy as compared with delayed BWL therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT + hormonal intensification). Measured by Cancer and Aging Research Group- Geriatric Assessment (CARG-GA) and Geriatric 8 (G8) instruments. T test will be used to compare CARG-GA and G8 change scores between two arms (T2 [3 month after treatment initiation] minus T1 [before or at treatment initiation]).
Difference in overall quality of life | Baseline to 3 months post ADT combination treatment initiation
  Will compare the difference in overall quality of life between men with prostate cancer receiving immediate BWL therapy as compared with delayed BWL therapy during ADT combination treatment (ADT + chemotherapy + hormonal intensification OR ADT + hormonal intensification). Measured by Functional Assessment of Cancer Therapy (FACT)-Prostate (FACT-P) instrument. T test will be used to compare FACT-P change score between two arms (T2 [3 month after treatment initiation] minus T1 [before or at treatment initiation]).

CONTACTS AND LOCATIONS:
Overall Officials: William Dale, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States